CLINICAL TRIAL: NCT00771147
Title: Prospective Open-label Non-interventional, Non-controlled Multi Observational and Pharmaco-economic Phase IV Trial to Evaluate the Characteristics of Patients Treated for Advanced Renal Cell Carcinoma With Nexavar ® as Well as Effectiveness, Safety and Direct Medical Costs of Nexavar® Treatment Under Daily-life Treatment Conditions
Brief Title: A Trial to Evaluate the Characteristics of Patients Treated for Advanced Renal Cell Carcinoma With Nexavar ®
Acronym: PONDIAC
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer Healthcare AG
Other Study IDs: 13102; NX0710BE
Record Dates: First submitted 2008-10-09; First posted 2008-10-13 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Carcinoma, Renal Cell; Carcinoma, Renal Cell (Advanced)
Keywords: Advanced Renal Cell Carcinoma ( RCC)
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Patients with diagnosis of advanced renal cell cancer and decision taken by the investigator to prescribe Nexavar®.

SUMMARY:
Evaluation of the efficacy and safety of Nexavar ® in advanced Renal Cell Carcinoma (RCC) and calculation of related medical costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of advanced RCC and decision taken by the investigator to prescribe Nexavar®. The patients should have sufficient knowledge of French or Dutch to be able to participate in the Study

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the Belgian product information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of advanced Renal Cell Carcimona
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2008-06; Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are progression-free at one year according to the RECIST criteria. The proportion of patients who are progression-free at 1, 3, 6 and 9 months will also be calculated | At 1, 3, 6 and 9 months and after one year

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Belgium